CLINICAL TRIAL: NCT06675461
Title: Randomized Controlled Trial of a Brief Psychological Intervention for Suicidal Patients With Borderline Personality Disorder in the Emergency Department
Brief Title: Brief Psychological Intervention for Suicidal Patients With Borderline Personality Disorder in the Emergency Department
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Anne Sonley, Associated Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-081
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: Brief Intervention; Brief Treatment; Treatment; Intervention; Gold Card
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Active Comparator): Access to psychiatric assessment, medication review, and unscheduled sessions with allied health professionals using a drop-in model of care.
  Interventions: Behavioral: Treatment as usual
- Gold Card Intervention (Experimental): A 4-session manualized intervention consisting of weekly scheduled 50-minute 1:1 sessions focused on psycho-education, here-and-now problem solving and safety planning. One of the sessions can involve a significant other to provide psychoeducation about the disorder and to facilitate support.
  Interventions: Behavioral: Gold Card Intervention

INTERVENTIONS:
Behavioral: Gold Card Intervention — A 4-session manualized intervention consisting of weekly scheduled 50-minute 1:1 sessions focused on psycho-education, here-and-now problem solving and safety planning. One of the sessions can involve a significant other to provide psychoeducation about the disorder and to facilitate support.
  Arms: Gold Card Intervention
Behavioral: Treatment as usual — Access to psychiatric assessment, medication review, and unscheduled sessions with allied health professionals using a drop-in model of care.
  Arms: Treatment As Usual

SUMMARY:
When in crisis, people with borderline personality disorder (BPD) frequently seek care in emergency departments (EDs) often presenting with suicide and self-harm behaviour. There is no established evidence-based brief treatment for patients with BPD in ED settings, however a 4-session treatment for people with personality disorders in ED settings was tested in Australia and showed promising results in reducing health care use and improving symptoms. A recent pilot feasibility randomized controlled trial (RCT) comparing this 4-session treatment to treatment as usual was conducted at the Centre for Addiction and Mental Health and preliminary findings have shown that the treatment is feasible to deliver and acceptable to both patients and clinicians. The proposed fully powered RCT will build on this pilot data to assess the efficacy of delivering this 4-session intervention in the ED for people with BPD who present with suicidal ideation or self-harm with the aim of reducing emergency health care use and improving BPD symptoms, functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have capacity to provide informed consent;
2. Must sign and date the informed consent form;
3. Stated willingness to comply with all study procedures;
4. Aged 16 or older;
5. Presenting to ED with self-harm and/or suicidal ideation;
6. Meeting criteria for BPD on the International Personality Disorders Examination (IPDE).
7. Endorsing a score of 1 or greater on the Suicide Ideation Attributes Scale (SIDAS).

Exclusion Criteria:

1. Meeting DSM-5 criteria for schizophrenia spectrum disorder or bipolar disorder I mania based on the Structured Clinical Interview for DSM-5 (SCID-5);
2. Severe alcohol or substance use disorder based on the Structured Clinical Interview for DSM-5 (SCID-5) requiring medical detoxification or residential treatment.
3. IQ < 70 based on the Test of Premorbid Functioning (TOPF).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | 6 Month Follow Up
  Suicidal Ideation Attributes Scale (SIDAS): is a self-report questionnaire that assesses history and severity of suicidal behaviour and ideation. Scores range from 0-50 with lower scores indicating less suicidal ideation.

SECONDARY OUTCOMES:
Suicidal Ideation | 3 Month Follow Up
  Suicidal Ideation Attributes Scale (SIDAS): is a self-report questionnaire that assesses history and severity of suicidal behaviour and ideation. Scores range from 0-50 with lower scores indicating less suicidal ideation.
Health Care Use | 3 and 6 Month Follow Up
  Client Service Receipt Inventory (CSRI): is a brief self-report questionnaire assessing the frequency of patient contact with health, social care or other professionals, as well as emergency departments visits and hospital admissions.
Borderline Personality Disorder Symptoms | 3 and 6 Month Follow Up
  Borderline Symptom Checklist-23 (BSL-23): is a self report questionnaire that assesses BPD symptoms during the previous week. The 23-item questionnaire has patients rate their experience of symptoms on a 5-point scale from 0 (not at all) to 4 (very strong). Total score is an average with a minimum of 0 and a maximum of 4. Higher scores indicate more BPD symptoms.
Self-Harm Behavior | 3 and 6 Month Follow Up
  Deliberate Self-Harm Inventory (DSHI): is a 17-item self-report questionnaire measuring frequency, severity, duration, and type of self-harm, which is defined as the direct destruction of body tissue.
Emotion Regulation | 3 and 6 Month Follow Up
  Difficulties in Emotion Regulation Scale (DERS): ) is a self-report questionnaire that measures six facets of emotion regulation. Scores range from 0-180 with higher scores indicating more emotional dysregulation.
Depressive Symptoms | 3 and 6 Month Follow Up
  Patient Health Questionnaire-9 (PHQ-9): is a 9-item self-report questionnaire assessing depression severity. Scores range from 0-27 with higher scores indicating more severe depression.
Functioning | 3 and 6 Month Follow Up
  WHO Disability Assessment Schedule (WHODAS): is a self-report questionnaire measuring health and disability across all diseases, including mental, neurological and addictive disorders. It assesses functioning in cognition, mobility, self-care, getting along, life activities and participation. Total score can range from 0-100 with 100 indicating full disability.
Quality of Life | 3 and 6 Month Follow Up
  WHO Quality of Life (WHOQOL): is a brief self-report questionnaire assessing quality of life in domains of physical and psychological health, interpersonal relationships and environment. Scores range from 0-100 with 100 indicating the best possible state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No